CLINICAL TRIAL: NCT06163339
Title: Evaluation of the Cultural Formulation Interview (CFI) - An Interview Support Aiming to Enhance Assessment and Treatment Adherence
Brief Title: Evaluation of the Cultural Formulation Interview (CFI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Christina Dalman, Professor, Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: jaka01
Record Dates: First submitted 2023-11-15; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Mental Health Issue
MeSH Terms: interventions — chemotactic factor inactivator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CFI + Usual Care (Experimental): About half of participants who are allocated to a person who works with the CFI during the trial.
  Interventions: Other: Cultural Formulation Interview
- Usual Care (No Intervention): About half of participants who are allocated to a person who do not work with the CFI during the trial (i.e., usual care).

INTERVENTIONS:
Other: Cultural Formulation Interview — Usual Care is enhanced with the Cultural Formulation Interview (CFI) aimed at strengthening assessment and treatment adherence
  Other Names: CFI
  Arms: CFI + Usual Care

SUMMARY:
Studies show that the mental health of children may have deteriorated in recent decades. In Sweden, several national initiatives have been implemented to develop and strengthen interventions for children's mental health. One of these initiatives involves enhancing the first line of primary care for children with mental health issues, whose mission is to provide early intervention, i.e., support for mild to moderate mental health problems. The responsibility for children with moderate to severe mental health issues lies with child and adolescent psychiatry.

Research indicates that children with a migration background, to a lesser extent than native-born children, have contact with both the first line of mental health care and child and adolescent psychiatry. There is also research showing that when newly arrived individuals do seek care, they may receive poorer quality care than others and, for example, may be misunderstood. From the perspective of equal healthcare, this is a significant shortcoming. In our study, the investigators address differences between healthcare providers and families based on cultural factors as a possible reason for the lack of equality in healthcare.

In the study, the investigators aim to evaluate whether the Cultural Formulation Interview (CFI) improves the connection between healthcare providers and families and increases the family's involvement in treatment, ultimately leading to better mental health for the child. The method can be said to aim at enhancing the assessment, compliance, and treatment that are currently available within healthcare.

DETAILED DESCRIPTION:
The overall aim of the project is is to evaluate the effects and experiences of the CFI, which aims to be a tool for assessing mental health regardless of cultural background. Developed by world-leading researchers in the field, CFI is intended to support psychiatric diagnosis, strengthen the alliance between healthcare providers and patients, and contribute to treatment planning that both parties agree on, thereby increasing adherence to treatment.

The specific research questions are:

Study Part 1 (Quantitative Method):

1. Do caregivers, where the child undergoes an enhanced assessment with CFI (i.e., standard care + CFI), report better working alliance and treatment credibility compared to children receiving standard care?
2. Do caregivers, where the child undergoes an enhanced assessment with CFI, report reduced mental health issues and increased quality of life compared to children receiving standard care?

Study Part 2 (Qualitative Method):

1. How do caregivers experience the CFI interview questions and the assessment conversation with the healthcare provider?
2. Do caregivers' gender and background factors (such as country of birth, migration experience, socioeconomic conditions, and occupation) influence their perception of CFI?
3. How do caregivers perceive the child's reaction to CFI and the assessment conversation?
4. How does CFI impact caregivers' understanding of healthcare and their sense of involvement?
5. What is the staff's experience with CFI? (For example, regarding understanding the patient's difficulties, perspectives on illness, and socio-cultural context).
6. How does CFI affect staff's interactions with patients and families?
7. How do staff perceive the practical feasibility of CFI? (For example, in terms of time commitment and documentation).
8. How do staff perceive that information from CFI influences the diagnosis, assessment, and treatment of healthcare needs?

CFI is developed by leading researchers in the field and is a tool intended to support psychiatric diagnosis, strengthen the alliance between healthcare providers and patients, and contribute to treatment planning that both parties agree on, thereby increasing adherence. The main interview consists of 16 open-ended questions that explore the patient's perspectives and context, including how social and cultural factors can influence expressions, explanatory models, coping strategies, and expectations of healthcare. The interview can be used by various professional categories such as physicians, psychologists, and counselors, and there is flexibility for healthcare providers to reformulate and choose questions they deem relevant for the assessment. The interview is intended for all patients but may be particularly useful in transcultural encounters. In addition to the main interview, there is also an interview targeting family members, as well as 12 in-depth supplementary modules. , one of which is designed for school-age children and adolescents and their parents.

Study Part 1 (Quantitative Method):

Healthcare providers (i.e., psychologists or counselors) at the participating clinics (Region Stockholm) will be randomly assigned to whether they will work with CFI during the study or not. Those working with CFI will receive training in the method before the study begins. Patients are referred to healthcare providers according to the clinic's procedures, often involving the provider with the shortest waiting time. To evaluate the effect of CFI on treatment credibility, working alliance with the healthcare provider, and the child's mental health, reliability and validity-tested rating scales will be used.

Study Part 2 (Qualitative Method):

Among the caregivers who participated in the assessment with CFI, some (approximately 10-15 individuals) will be interviewed, focusing on their experiences with CFI and their interactions with the clinic. Also, the staff who worked with CFI will be interviewed individually or in focus groups regarding their experience with CFI (n=5). These interviews (with caregivers and staff) will be conducted by members of the EPiCSS research group (Karolinska Institutet) using semi-structured interview guides based on themes. Interviews with caregivers and staff are offered on-site at the clinic or via phone or Zoom, conducted in Swedish or, if necessary, in English or through an interpreter.

Study Part 1 (Quantitative Method):

Within two-three weeks after the assessment interview (CFI interview or a corresponding visit in the control group), online survey data are collected regarding caregivers' confidence that the intervention their child will be offered at the clinic will help them (i.e., treatment credibility).

Three months after the CFI or corresponding visit, another online survey is sent to parents. The survey collects data on caregivers' experience of collaboration with the healthcare provider (i.e., working alliance) and caregivers' ratings of the child's mental health.

Study Part 2 (Qualitative Method):

Interviews about caregivers' experiences with CFI take place within three weeks after the caregiver has been interviewed with CFI. Interviews with staff occur at the earliest a couple of months after staff members start using CFI. The audio from interviews (both for caregivers and staff) regarding the experience of CFI is recorded.

ELIGIBILITY:
Inclusion Criteria:

Study Part

* Children between the ages of 6-14
* Families seeking care at any of the participating clinics
* Families assessed as suitable for interventions at the clinic where they seek care.

Study Part 2

* Caregivers who have consented to participate in Part 1 and have been interviewed using CFI as part of the study
* Healthcare providers/personnel who have used CFI as part of Part 1.

Exclusion Criteria:

Study Part 1

* Children who have not yet turned 6 years old and individuals aged 15 and above
* The child is assessed as not suitable for interventions at the clinic where they seek care.

Study Part 2

* Caregivers who have not consented to participate in Part 1.
* Caregivers who have not been interviewed using CFI as part of the study.
* Healthcare providers/personnel who have not used CFI as part of Part 1.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 248 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Credibility Scale | Two-three weeks after the baseline assessment
  The scale includes four statements (for example, "So far, how well do you think this care seems to fit your problems?"). The informant can respond on a Likert scale ranging from 0 to 10.

SECONDARY OUTCOMES:
KIDSCREEN-10 | Three months after the baseline assessment
  The scale aims to measure the child's well-being and includes 10 statements (for example, "Thinking about last week... did your child feel full of energy?"). The caregiver responds on a Likert scale with five options ranging from "Never" to "Always."
The Revised Child Anxiety and Depression Scale | Three months after the baseline assessment
  The scale aims to jointly measure the child's anxiety and depression symptoms, and consists of 25 statements (for example, 'My child worries about things') where the caregiver responds on a Likert scale with four options ranging from 'Never' to 'Always. The sum of all 25 items represent a broad measure of internalized symptoms.
Working Alliance Inventory | Three months after the baseline assessment
  The scale consists of six statements (for example, "Our therapist and we worked towards mutually agreed-upon goals") where the informant can respond using a Likert scale with six options ranging from "Not at all" to "Completely."

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dalman, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Solna, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data may be shared, given that it is possible due to legislation in Sweden